CLINICAL TRIAL: NCT04723199
Title: Feasibility of EUS-guided Biliary Drainage With a New-type of Eletrocautery LAMS for the Treatmentof Patients With Distal Malignant Biliary Obstruction (SPAZUS)
Brief Title: Feasibility of EUS-guided Biliary Drainage With LAMS for the Treatmentof Patients With Distal Malignant Biliary Obstruction
Acronym: SPAXUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 102
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Biliary Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrocautetery LAMS — Electrocautetery LAMS

SUMMARY:
Distal malignant biliary obstruction results from different types of tumors including pancreatic cancer, biliary tract cancer (BTC), gallbladder cancer, and metastasis, which can lead to obstructive jaundice. Endoscopic retrograde cholangiopancreatography (ERCP) represents the gold standard for jaundice palliation in this setting of patients. However, surgically altered anatomy (i.e., Whipple intervention, Roux-en-Y gastric bypass, Billroth II surgery), periampullary diverticula, gastric outlet obstruction, and malignant obstruction of the lumen determine the failure of the procedure in about 5-10% of cases, requiring alternative methods of decompression. Percutaneous transhepatic biliary drainage (PTBD) and surgical bypass are well established alternatives in these patients, but associated with increased morbidity, longer length of hospital stay and higher costs, and patient discomfort.

In 2001 Giovannini et al. described the first EUS guided biliary drainage (EUS-BD) through a transduodenal access with a needle knife.

Subsequently, EUS-BD has considerably evolved thanks to the development of dedicated devices such as lumen apposing metal stents (LAMS), specifically designed for endoscopic ultrasound procedures. LAMS are made up of braided nitinol, that is fully covered with silicone to prevent tissue ingrowth, with wide flanges on both ends to provide anchorage.

Recently, LAMS have been incorporated into a delivery system with an electrocautery mounted on the tip (Hot Axios; Boston Scientific Corp.), which allows the device to be used directly to penetrate the target structure without the need to utilize a 19G needle, a guidewire, and a cystotome for prior dilation. This has been described for drainage of peri-pancreatic fluid collections, common bile duct (CBD), gallbladder, and for creation of gastro-jejuno anastomosis. The biliary drainage procedure performed with the Hot Axios sistem is a one step procedure that requires less or no need for accessory exchange and becomes faster, thus potentially decreasing the risk of complications.

The procedure has been described as safe and effective with a technical success of 98.2 %, clinical success of 96.4 %, and low rate of complications 7 % (duodenal perforations, bleeding and transient cholangitis). A systematic review and meta-analyses showed clinical and technical success rates of 87% and 95% respectively. Currently, the EUS-BD is indicated as a rescue therapy for jaundice palliation after ERCP failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with distal malignant biliary obstruction
* Dilated common bile duct (>15 mm diameter) at either abdominal ultrasound, computed tomography, magnetic resonance or EUS or accessible gallbladder from the duodenum or from the stomach for the drainage
* Agree to receive follow up phone calls
* Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders and/or INR>1.5, PLT<50,000
* Use of anticoagulants that cannot be discontinued
* Pregnant women
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational multicentric prospective study coordinated by Dr. Benedetto Mangiavillano, Gastroenterology and Gastrointestinal Endoscopy Unit, Humanitas Mater Domini, Castellanza (VA), Italy. Data from consecutive patients with jaundice caused by distal malignant biliary obstruction will be evaluated and, if eligible and agreed to participate, will be recorded in an electronic register. Patients will be followed until death or for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of technical success | 12 Months
  The rate of successful LAMS placement in the targeted organ
Rate of clinical success | 12 Months
  Decrease of the total bilirubin levels > 20% at 24 hours after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Mater Domini, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No